CLINICAL TRIAL: NCT02792751
Title: Effects of Bispectral Index on Oxidative Stress
Brief Title: Does the Use of Bispectral Index Reduce the Oxidative Stress in Endoscopic Retrograde Cholangiopancreatography?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 123
Record Dates: First submitted 2016-05-27; First posted 2016-06-08 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-05

CONDITIONS: Oxidative Stress
Keywords: Depth of anesthesia; BIS; ERCP; Positive Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group R (Ramsey)=25 patients (Active Comparator): Propofol infusion was administered to provide Ramsey Sedation Scale 3-4 in Group R
  Interventions: Other: Ramsey Sedation Scale
- Group B (BIS)=25 patients (Experimental): Propofol infusion was given to maintain the Bispectral index monitorisation (BIS) levels between 60 and 85 in Group B.
  Interventions: Device: Bispectral Index Monitorisation (BIS)

INTERVENTIONS:
Device: Bispectral Index Monitorisation (BIS) — Standard monitoring was performed with electrocardiography, pulse oximetry and non invasive blood pressure. Additionally, Bispectral index (Aspect Medical Systems, Natica, MA) electrodes were connected to Group B patients
  Arms: Group B (BIS)=25 patients
Other: Ramsey Sedation Scale — Propofol administration was done to keep the Ramsey Sedation scale of 3 or 4
  Arms: Group R (Ramsey)=25 patients

SUMMARY:
Objective Endoscopic Retrograde Cholangiopancreatography (ERCP) is performed for resolving cholestasis by sphincterotomy and/or stone extraction and is done with deep sedation or general anesthesia. The investigators primary outcome was to evaluate the effects of the depth of anesthesia on oxidative stres provided via Bispectral Index (BIS) monitorisation during the ERCP procedure by analyzing the biochemical parameters. And their secondary outcome was the effects of anesthesia depth on propofol consumption and postoperative sedation status.

DETAILED DESCRIPTION:
50 patients undergoing ERCP procedure were randomly allocated in two groups. Propofol was given to provide the patients Ramsey sedation scale as 3 and 4 in Group R (n=25) patients whereas it was given to Group B (n=25) patients to provide BIS values between 65 to 85. The levels of total oxidant status (TOS), total antioxidant status (TAS), and Oxidative stres index (OSI) were measured. Hemodynamic signs, propofol consumption, postoperative recovery time were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status I-II
* Patients undergoing ERCP procedures

Exclusion Criteria:

* uncontrolled comorbidities (hypertension, diabetes mellitus, kidney-liver failure)
* difficulty in communication (language problems, such as deafness)
* who are allergic to the drugs used
* pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effects of BIS on oxidative stress | one day
  The investigators aimed to investigate the effects of anesthesia with monitoring the depth of anesthesia using BIS on oxidative stres by measuring the total oxidant status (TAS) and total antioxidant status (TOS) , propofol consumption, and postoperative recovery during ERCP procedures in this study.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data